CLINICAL TRIAL: NCT06369558
Title: Effectiveness of Plyometric Exercise Training in Athletes With Chronic Low Back Pain: A Randomized Controlled Trial
Brief Title: Plyometric Exercise Training in Athletes With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ugur Cavlak (Other)
Collaborators: Biruni University (Other)
Responsible Party: Sponsor-Investigator, Ugur Cavlak, CLINICAL PROFESSOR, Biruni University
Organization: Biruni University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BiruniUniversi
Record Dates: First submitted 2024-04-04; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Low Back Pain, Mechanical
Keywords: Chronic Low Pain; Plyometric exercise; Physiotherapy; Athlete
MeSH Terms: conditions — Low Back Pain | interventions — Plyometric Exercise

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PYLOMETRIC (Experimental): PLYOMETRIC TRAINING
  Interventions: Other: PLYOMETRIC TRAINING
- CONTROL (Active Comparator): CLASSIC PHYSIOTHERAPY PROGRAM
  Interventions: Other: PLYOMETRIC TRAINING; Other: CLASSIC PHYSIOTHERAPY PROGRAM

INTERVENTIONS:
Other: PLYOMETRIC TRAINING — A 6 WEEK (3 TIMES A WEEK) CONSISTING OF JUMPING SINGLE LEG BRIDGE AND JUMPED SQUAT
Other: CLASSIC PHYSIOTHERAPY PROGRAM — HOT PACKED ENTEFERANTIAL CURRENT THERAPY AND US THERAPY
  Arms: CONTROL

SUMMARY:
The aim of this study is to examine the effectiveness of plyometric exercise training in the athletes with chronic low back pain. 32 professional volunteer athletes participated in the study.

DETAILED DESCRIPTION:
Visual Analog Scale (VAS) for pain assessment and Oswestry Disability Index for disability level will be used. Sit and Reach Test, Vertical Jump, Flamingo balance test and Shuttle Running test (20 min.) will be used to measure the physical functioning of the participants. Manual Muscle testing will also be used to measure the participants' lower and upper muscles. The participants were divided into two groups. The interventional program will be finished after 6 weeks (3 days a week). The program includes; physical therapy session (Hot packed, vacuum interferential current therapy, therapeutic ultrasound, exercises) and plyometric exercises.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-25
* Being a licensed athlete (male of famele)
* Low back pain is chronic and lasts at least 3 months

Exclusion Criteria:

* Having had back pain or any surgery that caused it in the last year.
* Having cardiovaskular disease
* Doping and using banned substances.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
VISUAL ANALOG SCALE | baseline and immediately after the intervention
  TO MEASURE PAIN INTENSITY (MİN.-MAX.:0-10 POINT)
OSWESTRY DISABILITY INDEX | baseline and immediately after the intervention
  TO MEASURE PAIN DISABILITY (MİN.-MAX.:0-50 POİNT)
SIT AND REACH TEST | baseline and immediately after the intervention
  TO MEASURE MUSCLE FLEXIBILITY (MİN.-MAX.:0-29 POİNT)
VERTICAL JUMP TEST | baseline and immediately after the intervention
  EXPECT TO HİGER SCOE İN CENTIMETER
FLAMINGO BALANCE TEST | baseline and immediately after the intervention
  TO MEASURE BALANCE (MİN.-MAX.:0-60 SECOND)
SHUTTLE RUNNİNG (20 MİN.) | baseline and immediately after the intervention
  TO MEASURE FUNCTIONALITY
MANUAL MUSCLE STRENGTH TEST | baseline and immediately after the intervention
  TO MEASURE MUSCLE STRENGTH

CONTACTS AND LOCATIONS:
Overall Officials: UGUR CAVLAK, Principal Investigator — Biruni University
Locations (1):
- Faculty of Health Sciences in Biruni University, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huang PY, Jankaew A, Lin CF. Effects of Plyometric and Balance Training on Neuromuscular Control of Recreational Athletes with Functional Ankle Instability: A Randomized Controlled Laboratory Study. Int J Environ Res Public Health. 2021 May 15;18(10):5269. doi: 10.3390/ijerph18105269. PMID 34063454